CLINICAL TRIAL: NCT05505357
Title: Omission of Breast Surgery for Predicted Pathologic Complete Response Patients With MRI and Vacuum-assisted bIopsy in Breast Cancer After Neoadjuvant Systemic Therapy: a Multicenter, Single-arm, Non-inferiority Trial
Brief Title: Omission of Breast Surgery for Breast Cancer Patients With pCR on MRI and Vacuum-assisted Biopsy After NST (OPTIMIST)
Acronym: OPTIMIST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ministry of Health & Welfare, Korea (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KBCSG-24
Record Dates: First submitted 2022-08-16; First posted 2022-08-17 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer Invasive
Keywords: neoadjuvant systemic therapy; pathological complete response; vacuum-assisted bIopsy; omission of breast surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with pCR predicted by MRI and vacuum-assisted biopsy (VAB) after neoadjuvant chemotherapy (Experimental): When there is no residual tumor cells on the vacuum-assisted biopsy specimen, breast surgery will be omitted. In the case of clinical N0 AND MRI size ≤ 0.5cm AND lesion-to-background signal enhancement ratio ≤1.6, sentinel lymph node biopsy will be omitted. Otherwise, sentinel lymph node biopsy will be performed. If necessary, axillary lymph node dissection will be performed.
  Interventions: Procedure: Breast surgery omission

INTERVENTIONS:
Procedure: Breast surgery omission — For patients who are expected to achieve pathologic complete response after neoadjuvant chemotherapy based on MRI findings, vacuum-assisted biopsy will be performed on the main primary lesion marked with a clip. In case of pCR on vacuum-assisted biopsy specimen, breast surgery will be omitted.

SUMMARY:
A prospective, multicenter, single-arm non-inferiority trial to demonstrate that breast cancer patients who are predicted to have a pathologic complete response on MRI and vacuum-assisted biopsy after neoadjuvant systemic therapy, and are omitted breast surgery have a non-inferior 5-year disease-free survival compared to those who had received breast surgery.

DETAILED DESCRIPTION:
[Background & Rationale for Study]

Optimization (rather than de-escalation) of surgery for breast cancer is essential for our patients, and thus it is an important topic discussed actively in all major conferences regarding breast cancer and oncology.

A previous study showed that lesion-to-background parenchymal signal enhancement ratio (L-to-B SER) ≤1.6 and/or size ≤ 0.2cm on breast MRI can distinguish pathological complete response (pCR) from minimal residual cancer following neoadjuvant systemic therapy (NST). In a separate prospective study, 40 patients with near pCR (either tumor size ≤ 0.5 cm or L-to-B SER ≤ 1.6 on MRI) were enrolled and evaluated for the accuracy of US-guided biopsy aided by MRI in predicting pCR in the breast after NST. US-guided multiple core needle biopsy (CNB) or VAB of the tumor bed, followed by standard surgical excision, was performed. Matched biopsy and surgical specimens were compared to assess pCR. In result, obtaining at least 5 biopsy cores based on tumor size ≤ 0.5 cm and an L-to-B SER of ≤ 1.6 on MRI resulted in 100% NPV and accuracy. No differences in accuracy were noted between CNB and VAB (90% vs. 90%). It was demonstrated that patients who meet these stringent criteria on MRI may forego surgery for breast cancer.

Also, a pooled analysis of data from The Royal Marsden, MD Anderson Cancer Center, and Seoul National University Hospital showed that a VAB obtaining at least 6 cores for a lesion ≤2cm on imaging after NST can accurately predict pCR at a FNR of 3.2%.

For patients who would not benefit from surgery, it is unnecessary in terms of both personal and national medical expenses. Therefore, in order to establish the rationale for whether surgery could be omitted for patients with predicted pCR, it is necessary to demonstrate that the survival rate of patients who skipped breast surgery after confirming no residual cancer on VAB is non-inferior than that of patients who underwent breast surgery.

[Study Objectives]

To show non-inferiority in terms of disease-free survival (DFS) of omission of breast surgery for breast cancer patients who show no residual tumor on VAB after NST.

[Study design]

Prospective, multicenter, single-arm, non-inferiority trial

ELIGIBILITY:
Inclusion Criteria:

* Sex: female
* Age: 20 years and older
* Patients with no clinical/radiologic distant metastasis
* Tumor type: Invasive ductal carcinoma
* Tumor subtype: HER2 positive(including luminal B type, triple negative
* Extent of disease: initial tumor size ≤ 5cm, cN0-2
* Patients with measurable tumor size
* Patients who are expected to achieve pCR after neoadjuvant chemotherapy (MRI size ≤ 1.0 cm AND L-to-B SER ≤ 1.6)
* Patients with clip inserted to the primary tumor site before or during neoadjuvant chemotherapy
* Patients with informed consent who are competent to make a voluntary decision

Exclusion Criteria:

* Multifocal lesion (≥2)
* Extent of residual microcalcification after neoadjuvant chemotherapy > 2cm
* Bilateral breast cancer or inflammatory breast cancer
* Contraindication to radiotherapy
* History of previous contralateral breast cancer
* Breast cancer patients with distant metastasis
* Allergic history to MRI contrast
* Male breast cancer
* Patients incapable of giving informed consent owing to poor general conditions
* Patients with BRCA mutation
* Patients willing to receive breast surgery
* Patients with a history of cancer diagnosis within 5 years (However, skin cancer other than melanoma and breast carcinoma in situ other than ductal carcinoma in situ can be registered even if 5 years have not passed since the diagnosis)

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 533 (Estimated)
Dates: Start 2022-09-22 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival | 5 years after axillary surgery or VAB (in case of axillary surgery omission)
  Proportion of patients with no disease recurrence (including loco-regional recurrence, distant metastasis, and contralateral breast cancer) or death.

SECONDARY OUTCOMES:
Ipsilateral Breast Tumor Recurrence-Free Survival Ipsilateral Breast Tumor Recurrence-Free Survival | 5 years after axillary surgery or VAB (in case of axillary surgery omission)
  Proportion of patients with no disease recurrence in the ipsilateral breast or death
Overall Survival | 5 years after axillary surgery or VAB (in case of axillary surgery omission)
  Proportion of patients with no death.
Invasive Disease-Free Survival Invasive Disease-Free Survival | 5 years after axillary surgery or VAB (in case of axillary surgery omission)
  Proportion of patients with no invasive disease recurrence (including loco-regional recurrence, distant metastasis, and contralateral breast cancer) or death.
QoL, symptoms, and medical cost | 1 year after axillary surgery or VAB (in case of axillary surgery omission)
  Analysis of QoL survey (BREAST-Q), procedure-related symptoms, and medical cost
Rate of residual axillary lymph node metastasis on axillary surgery | Upon axillary surgery
  Proportion of patients with metastatic lymph nodes among those with pCR on VAB

CONTACTS AND LOCATIONS:
Overall Officials: Han-Byoel Lee, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Available on Request (hblee80@gmail.com; hblee.md@snu.ac.kr)
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: March 2032
Access Criteria: Upon request

REFERENCES:
- [Background] Kim SY, Cho N, Shin SU, Lee HB, Han W, Park IA, Kwon BR, Kim SY, Lee SH, Chang JM, Moon WK. Contrast-enhanced MRI after neoadjuvant chemotherapy of breast cancer: lesion-to-background parenchymal signal enhancement ratio for discriminating pathological complete response from minimal residual tumour. Eur Radiol. 2018 Jul;28(7):2986-2995. doi: 10.1007/s00330-017-5251-8. Epub 2018 Jan 29. PMID 29380033
- [Background] Lee HB, Han W, Kim SY, Cho N, Kim KE, Park JH, Ju YW, Lee ES, Lim SJ, Kim JH, Ryu HS, Lee DW, Kim M, Kim TY, Lee KH, Shin SU, Lee SH, Chang JM, Moon HG, Im SA, Moon WK, Park IA, Noh DY. Prediction of pathologic complete response using image-guided biopsy after neoadjuvant chemotherapy in breast cancer patients selected based on MRI findings: a prospective feasibility trial. Breast Cancer Res Treat. 2020 Jul;182(1):97-105. doi: 10.1007/s10549-020-05678-3. Epub 2020 May 16. PMID 32418044
- [Background] Tasoulis MK, Lee HB, Yang W, Pope R, Krishnamurthy S, Kim SY, Cho N, Teoh V, Rauch GM, Smith BD, Valero V, Mohammed K, Han W, MacNeill F, Kuerer HM. Accuracy of Post-Neoadjuvant Chemotherapy Image-Guided Breast Biopsy to Predict Residual Cancer. JAMA Surg. 2020 Dec 1;155(12):e204103. doi: 10.1001/jamasurg.2020.4103. Epub 2020 Dec 16. PMID 33026457
- [Derived] Jung JJ, Cheun JH, Kim SY, Koh J, Ryu JM, Yoo TK, Shin HC, Ahn SG, Park S, Lim W, Nam SE, Park MH, Kim KS, Kang T, Lee J, Youn HJ, Kim YS, Yoon CI, Kim HK, Moon HG, Han W, Cho N, Kim MK, Lee HB. Omission of Breast Surgery in Predicted Pathologic Complete Response after Neoadjuvant Systemic Therapy: A Multicenter, Single-Arm, Non-inferiority Trial. J Breast Cancer. 2024 Feb;27(1):61-71. doi: 10.4048/jbc.2023.0265. PMID 38433091